CLINICAL TRIAL: NCT03397914
Title: Effect of Different Colistin Doses on Clinical Outcome of Pediatric Cancer Patients With Gram Negative Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Gram-Negative Bacterial Infections; Pediatric Cancer; Colistin; Colistin Adverse Reaction; MIC
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Neoplasms | interventions — colistinmethanesulfonic acid; Colistin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Regimen (Experimental): Randomized 30 pediatric subjects suffering from febrile neutropenia with proven or suspected gram negative infection will receive 2.5 mg/kg of colistimethate sodium intravenous as loading dose followed by 1.25 mg/kg every 12 hours as maintenance dose
  Interventions: Drug: Colistimethate Sodium
- Group B Regimen (Experimental): Randomized 30 pediatric subjects suffering from febrile neutropenia with proven or suspected gram negative infection will receive 5 mg/kg of colistimethate sodium intravenous as loading dose followed by 2.5 mg/kg every 12 hours as maintenance dose
  Interventions: Drug: Colistimethate Sodium

INTERVENTIONS:
Drug: Colistimethate Sodium — Intravenous injection of colistimethate Sodium 2.5 mg/kg or 5 mg/kg for Multidrug-resistance gram negative infections
  Other Names: Colimycin; Colistin Sulfate; Coly-Mycin; Polymyxin E

SUMMARY:
Prospective randomized study comparing different colistin dosing regimens in paediatric cancer patient with MDR gram-negative infection or sepsis

DETAILED DESCRIPTION:
The aim of this study is to:

1. Evaluate the clinical outcome of two different dosing regimen of IV colistin in the treatment of children with multidrug resistant gram-negative infections or sepsis.
2. To estimate the frequency of colistin associated adverse effects.
3. To correlate the serum colistin concentration and MIC to microbiological clearance and clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Age between one year and 18 years
2. All paediatric cancer patients who are prescribed intravenous colistin due to:

   * Sepsis due to MDR or minimally susceptible gram-negative bacteria
   * History of MDR gram-negative infection or sepsis due to organisms sensitive to colistin.
   * Culture result consistent with MDR gram negative for this febrile neutropenic episode.
   * Patient in sepsis and colistin was administered empirically to increase antibiotic coverage.

Exclusion Criteria:

1. Age less than one year or over 18 years
2. Patients with renal impairment
3. Colistin use less than 72 hours

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
clinical improvement, | 7- 14 days
  time to defervescence

SECONDARY OUTCOMES:
adverse events | 14 days
  incidence of colistin related nephropathy
microbiological clearance | 7-14 days
  time to clearance of cultures

CONTACTS AND LOCATIONS:
Overall Officials: Yosr Samia Abou Sedira, Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- Iman Sidhom, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storm DR, Rosenthal KS, Swanson PE. Polymyxin and related peptide antibiotics. Annu Rev Biochem. 1977;46:723-63. doi: 10.1146/annurev.bi.46.070177.003451. PMID 197881
- [Background] Komura S, Kurahashi K. Partial purification and properties of L-2,4-diaminobutyric acid activating enzyme from a polymyxin E producing organism. J Biochem. 1979 Oct;86(4):1013-21. doi: 10.1093/oxfordjournals.jbchem.a132594. PMID 500578
- [Background] Brown JM, Dorman DC, Roy LP. Acute renal failure due to overdosage of colistin. Med J Aust. 1970 Nov 14;2(20):923-4. doi: 10.5694/j.1326-5377.1970.tb63262.x. No abstract available. PMID 5486295
- [Background] Falagas ME, Kasiakou SK. Colistin: the revival of polymyxins for the management of multidrug-resistant gram-negative bacterial infections. Clin Infect Dis. 2005 May 1;40(9):1333-41. doi: 10.1086/429323. Epub 2005 Mar 22. PMID 15825037
- [Background] Dalfino L, Puntillo F, Mosca A, Monno R, Spada ML, Coppolecchia S, Miragliotta G, Bruno F, Brienza N. High-dose, extended-interval colistin administration in critically ill patients: is this the right dosing strategy? A preliminary study. Clin Infect Dis. 2012 Jun;54(12):1720-6. doi: 10.1093/cid/cis286. Epub 2012 Mar 15. PMID 22423120
- [Background] Hernandez Orozco H, Lucas Resendiz E, Castaneda JL, De Colsa A, Ramirez Mayans J, Johnson KM, Gonzalez N, Caniza MA. Surveillance of healthcare associated infections in pediatric cancer patients between 2004 and 2009 in a public pediatric hospital in Mexico city, Mexico. J Pediatr Hematol Oncol. 2014 Mar;36(2):96-8. doi: 10.1097/MPH.0b013e31827e7f4c. PMID 23337552
- [Background] Gupta A, Kapil A, Lodha R, Kabra SK, Sood S, Dhawan B, Das BK, Sreenivas V. Burden of healthcare-associated infections in a paediatric intensive care unit of a developing country: a single centre experience using active surveillance. J Hosp Infect. 2011 Aug;78(4):323-6. doi: 10.1016/j.jhin.2011.04.015. Epub 2011 Jun 14. PMID 21676495
- [Background] Bergen PJ, Li J, Nation RL. Dosing of colistin-back to basic PK/PD. Curr Opin Pharmacol. 2011 Oct;11(5):464-9. doi: 10.1016/j.coph.2011.07.004. Epub 2011 Aug 9. PMID 21835694